CLINICAL TRIAL: NCT02521597
Title: Mobile Otoscopy - Efficacy of Residents to Diagnose Acute Otitis Media Using a Smartphone Otoscope Attachment: A Randomized Controlled Trials
Brief Title: Mobile Otoscopy - Efficacy of Residents to Diagnose Acute Otitis Media Using a Smartphone Otoscope Attachment
Acronym: MOTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Jocelyn Gravel, MD, MSc, St. Justine's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: MOTO study
Record Dates: First submitted 2015-08-07; First posted 2015-08-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Acute Otitis Media
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cellscope (Experimental): The intervention for this study will be the use of a smartphone otoscope attachment called CellScope Oto.
  Interventions: Device: Cellscope
- Traditional otoscope (Active Comparator): The control group will be using a classic otoscope
  Interventions: Device: Traditional otoscope

INTERVENTIONS:
Device: Cellscope — The CellScope Oto, is a portable video-otoscope that allows residents and staff to share diagnostic-quality images
  Arms: Cellscope
Device: Traditional otoscope — Use of a regular otoscope
  Arms: Traditional otoscope

SUMMARY:
To evaluate the residents' efficacy in diagnosing acute otitis media among febrile children presenting with respiratory symptoms using a smartphone otoscope attachment compared with a classic otoscope.

DETAILED DESCRIPTION:
Background: Acute otitis media (AOM) is one of the most common diseases of childhood and a leading cause for health care consultations. While otoscope is the tool traditionally used to diagnose AOM, otoscopic diagnostic skills of both trainees and practitioners appear to be limited. Therefore, new diagnostic methods are continuously developed. One of those devices is a smartphone otoscope attachment called CellScope Oto, a portable video-otoscope that allows residents and staff to share diagnostic-quality images.

Objective: To evaluate the residents' efficacy in diagnosing acute otitis media among febrile children presenting with respiratory symptoms using a smartphone otoscope attachment compared with a classic otoscope.

Methods: This will be a randomized controlled trial evaluating accuracy of evaluation of ears of children visiting the emergency department (ED) for suspected AOM by residents using the CellScope Oto in comparison to a classic otoscope. It will be performed at a single pediatric ED in a tertiary care Hospital. Participants will be children between 1 and 5 years of age presenting with fever and respiratory symptoms. Baselines characteristics of participants will be assessed. Participating residents will be taught how to use the CellScope Oto and will practice with a few patients before being ready to participate in the study. Eligible patients will be recruited during weekdays. If the parents consent, patients will first be evaluated by a staff Pediatric Otolaryngologist using a binocular microscope (gold standard). They will then be evaluated by two participating residents, one using the intervention method and one using the control. Randomization will be used to decide which visualisation method will be used first. After all three exams have been performed, the residents, patients' parent and staff in charge will each be asked to answer a short questionnaire about final diagnosis and confidence in the performed exam, favourite method and the need for a control exam. These questionnaires will be reviewed by a reviewer blinded to the randomization. The primary outcome measure will be the accuracy of AOM diagnosis made by the residents compared with the diagnosis made by a staff Pediatric Otolaryngologist using a binocular microscope. A sample size of 100 participants evaluated twice would provide a power of 80% and an alpha value of 0,05 to demonstrate a difference of 15% in the rate of appropriate diagnosis of AOM by residents using a smartphone otoscope attachment compared with classic otoscope use.

Expected results: The investigators expect to demonstrate a 15% increase in the efficacy rate of AOM diagnosis by residents registered to a paediatrics-related program using a smartphone otoscope attachment compared with a classic otoscope. This device has the potential to change current AOM diagnostic practice and might, in turn, provide a reduced amount of prescriptions made every year for antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Visiting the ED for fever and respiratory problems
* During the hours when there is a research assistant

Exclusion Criteria:

* Anterior myringotomy with tube placement
* Signs of serious infection (triage priority 1 or 2, tachycardia and/or hypotension, bulging fontanelle, neck stiffness, purpuric rash, altered consciousness)
* Impossibility to obtain an informed consent by the parent (absence of parent, language barrier, etc)
* Severe chronic illness (immunodeficiency, congenital heart disease, encephalopathy, pulmonary disease other than asthma, and disorder of the ear, nose and throat)

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
accuracy in diagnosing acute otitis media | 15 minutes
  This will be the number of participants for which there will be a complete agreement between the evaluation of the resident and the diagnosis of acute otitis media as diagnosed by the Pediatric Otolaryngologist using binocular microscope.

SECONDARY OUTCOMES:
Need for second exam | 15 minutes
  The number of participants for which the staff in charge will have to repeat the exam
Parents satisfaction | 30 minutes
  The parents' satisfaction regarding the ear exam performed on their child using a likert scale
Confidence | 15 minutes
  the confidence of participants in their ear exams using a likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn Gravel, MD, MSc, Principal Investigator — St. Justine's Hospital
Locations (1):
- Sainte-Justine Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Mousseau S, Lapointe A, Gravel J. Diagnosing acute otitis media using a smartphone otoscope; a randomized controlled trial. Am J Emerg Med. 2018 Oct;36(10):1796-1801. doi: 10.1016/j.ajem.2018.01.093. Epub 2018 Jan 31. PMID 29544905